CLINICAL TRIAL: NCT03796208
Title: Behavioral and Enhanced Perinatal Intervention for Cessation (B-EPIC): Reducing Tobacco Use Among Opioid Addicted Women
Acronym: B-EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristin Ashford (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Kristin Ashford, Professor and Dean of Undergraduate Faculty Affairs, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45062; 1R34DA046005-01 (NIH)
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2021-12

CONDITIONS: Smoking Cessation
Keywords: Opioid Use Disorder; Pregnancy; tobacco
MeSH Terms: conditions — Smoking Cessation; Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobacco Intervention (Experimental): Participants in this group will be randomized to the Behavioral and Enhanced Perinatal Intervention for Cessation (B-EPIC) intervention.
  Interventions: Behavioral: Behavioral and Enhanced Perinatal Intervention for Cessation (B-EPIC)
- Treatment As Usual (Active Comparator): Participants in this group will be randomized to tobacco treatment as usual.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Behavioral and Enhanced Perinatal Intervention for Cessation (B-EPIC) — Women enrolled in the intervention group will receive TAU plus B-EPIC, which includes four core components: 1) Individualized tobacco treatment plus supplemental counseling, 2) Biomarker validation and feedback, 3) Change in maternal thought process and adoption of healthy behavior (e.g. exercise, based on PI framework), and 4) Pharmacotherapy as needed (see Table 3 for a summary of the study design). The initial assessment for this intervention takes 60 minutes, with follow-up sessions typically lasting 15-20 minutes. All sessions occur prior to or after pre-scheduled perinatal appointments. The intervention will be led by a certified tobacco treatment specialist (CTTS).
  Arms: Tobacco Intervention
Behavioral: Treatment As Usual — Women enrolled in the control group are informed of the risks of tobacco use and benefits of quitting using the ACOG 5'A's approach by their healthcare provider. This standard takes approximately 5-15 minutes, and is offered at each prenatal and postpartum appointment. The five steps of the ACOG recommendation are: 1.) Ask about tobacco use, 2.) Advise to quit, 3.) Assess willingness to make a quit attempt, 4.) Assist in quit attempt, and 5.) Arrange follow-up. The provider may also talk to the participant about nicotine replacement therapy.
  Arms: Treatment As Usual

SUMMARY:
This study tests an intervention for tobacco cessation (named B-EPIC) in an established community medication assisted treatment (MAT) clinic for pregnant and postpartum women with opioid dependence. Half of the participants will receive the intervention for tobacco cessation, which is standard cessation counseling from the provider plus additional cessation support from a Certified Tobacco Treatment Specialist (CTTS). The other half of participants will receive standard tobacco cessation from their provider. The project will also determine the economic impact of the B-EPIC intervention on healthcare expenditures.

DETAILED DESCRIPTION:
The study will use a prospective, 2-group, randomized, comparative effectiveness design to determine if the B-EPIC tobacco intervention is superior to tobacco 'treatment as usual (TAU)' for opioid dependent pregnant women maintained on buprenorphine; the outcomes for the first aim will be quitting smoking and/or reducing cigarette consumption during pregnancy. The project design also will determine the economic impact the B-EPIC intervention (10-months) has on healthcare expenditures.

After informed consent, eligible participants will be randomized (1:1) to the B-EPIC group (tobacco intervention) or TAU tobacco treatment (control group). All will continue to receive opioid dependence treatment with buprenorphine, regardless of treatment assignment.

Women enrolled in the control group are informed of the risks of tobacco use and benefits of quitting using the American College of Obstetricians and Gynecologists (ACOG) 5'A's approach by their healthcare provider. This standard tobacco cessation counseling takes approximately 5-15 minutes, and is offered at each prenatal and postpartum appointment.

Women enrolled in the intervention group will receive TAU plus B-EPIC, which includes four core components: 1) Individualized tobacco treatment plus supplemental counseling, 2) Biomarker validation and feedback, 3) Change in maternal thought process and adoption of healthy behavior (e.g. exercise, based on PI framework), and 4) Pharmacotherapy as needed. The initial assessment for this intervention takes 60 minutes, with follow-up sessions typically lasting 15-20 minutes. The intervention will be led by a certified tobacco treatment specialist (CTTS).

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of opioid dependence with participation in the University of Kentucky Healthcare and Baptist Health Lexington buprenorphine treatment program
* Less than 24 weeks gestation
* Age 18-49 years old
* Diagnosis of current tobacco use disorder
* Read or write in English

Exclusion Criteria:

* Current prisoner status
* Current severe mental illness (e.g., bipolar disorder with current mania, current suicidal ideation)
* Alcohol or sedative/hypnotic dependence that requires medical intervention

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All participants in this study will be pregnant females.
Enrollment: 78 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ashford, Principal Investigator — University of Kentucky; Amanda Fallin-Bennett, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Polk Dalton Clinic, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of individuals consented and further screened for eligibility = 79; Number of participants randomized to intervention = 40; Number of participants randomized to treatment as usual = 38
Pre-assignment Details: Participants may have been excluded prior to randomization for the following reason:
  1. Withdrawal (changed mind)
Period: Overall Study
Arm/Group | Tobacco Intervention | Treatment As Usual
Started | 40 | 38
Completed | 16 | 16
Not Completed | 24 | 22
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Loss of pregnancy | 1 | 1
Not completed — Changed prenatal clinics | 0 | 5
Not completed — Lost to Follow-up | 20 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobacco Intervention | Treatment As Usual | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 76
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.9 [22.7 to 43.5] | 30.8 [21.8 to 41.8] | 30.9 [21.8 to 43.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 33 | 35 | 68
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Cigarettes Smoked Per Day
Description: Participants will be asked during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks) to self-report the number of cigarettes smoked per day. Data will be presented as the change in the number of cigarettes smoked per day compared between groups.
Time Frame: up to 50 weeks (third trimester (28-36.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on number of participants with cigarettes smoked per day data available at third trimester (28-36.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change. Enrollment (up to 31.6 weeks gestation) was not used in this analysis due to a change in the data collection format from categorical to continuous. Disruptions by COVID-19 created many challenges with longitudinal data collection.
Measure: Median (Inter-Quartile Range); unit: cigarettes per day
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 15 | 18
cigarettes per day | 0 [-10 to 5] | 0 [-5 to 3]

2. Primary Outcome: Change in Urine Cotinine Concentration Level
Description: Participants will provide a urine sample to be measured by litmus analysis during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks). The litmus levels range from 0 (minimum) to 6 (maximum). Data will be presented as the change in cotinine levels by the litmus measure over the course of the study compared between groups.
Time Frame: up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with cotinine levels data available at enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change in the level of urine cotinine using NICALERT, an immunochromatographic assay test strip (Nymox Pharmaceutical Corporation, Montreal, Quebec). Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Mean (Standard Deviation); unit: litmus levels
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 22 | 24
litmus levels | -0.09 (0.68) | 0.17 (0.56)

3. Primary Outcome: Change in Electronic Cigarette Usage Per Day
Description: Participants will be asked during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks) to self-report electronic cigarette (e-cig) usage per day. Data will be presented as the change in e-cig usage per day compared between groups.
Time Frame: up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with self-report electronic cigarette (e-cig) usage per day and with data available at study time points enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change. Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Median (Inter-Quartile Range); unit: e-cig use times per day
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 4 | 6
e-cig use times per day | 1 [0 to 18] | -6 [-20 to 4]

4. Primary Outcome: Change in Cigarette Dependence
Description: Participants will complete the Fagerstrom Test for Cigarette Dependence during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks). The survey instrument asks seven questions related to cigarette dependency. For scoring, yes/no questions are scored from 0 to 1, and multiple choice questions from 0 to 3. Items are then summed to yield a total score of 0-10. The higher the total score, the more intense the patient's nicotine dependence. Any score greater than 8 is considered high dependency, a score of 5-7 is considered moderately dependent, 3-4 is low to moderate dependence and 1-2 is low dependence. Data will be presented as the change in cigarette dependency over time compared between groups.
Time Frame: up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with Fagerstrom Test for Cigarette Dependence data available at study time points enrollment (up to 31.6 weeks gestation) minus postpartum visit (2-8.6 weeks after delivery) to determine a change. Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 26 | 24
Score on a scale | 2.04 (3.14) | 1.42 (2.9)

5. Primary Outcome: Change in Electronic Cigarette Dependence
Description: Participants will complete the Penn State Electronic Cigarette Dependence Index (PSECDI) during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks). The survey instrument asks ten questions and responses are scored on a scale from zero to 20. Summed scores correlate to a dependence category; 0-3 is not dependent, 4-8 is low dependence, 9-12 is medium dependence, and above 12 is high dependence. Data will be presented as the change in electronic cigarette dependency over time compared between groups.
Time Frame: up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with Penn State Electronic Cigarette Dependence Index (PSECDI) data available at study time points enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change. Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 1 | 2
scores on a scale | -5.0 | -1.5 (2.12)

6. Secondary Outcome: Change in Maternal Depression Over Time
Description: Participants will complete the Edinburgh Postnatal Depression Scale (EPDS) during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks). The survey consisted of 10 multiple choice questions with scores for each question ranging from 0-3. Scores are then summed for a total score, ranging from 0-30. Questions 1, 2 & 4 are scored 0-3 with the first answer to each question scored as 0 and the fourth answer scored as 3. Questions 3 & 5-10 are reverse scored, with the first answer to each question scored as 3 and the fourth answer scored as 0. A score of 10 or greater is interpreted as "possible depression". A score of greater than 0 on item 10 indicates "suicidal thoughts". Data will be presented as the change in depression over time compared between groups.
Time Frame: Up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with Edinburgh Postnatal Depression Scale (EPDS) data available at study time points enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change. Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 26 | 26
score on a scale | 2.42 (3.86) | 2.58 (5.64)

7. Secondary Outcome: Change in Maternal Anxiety Over Time
Description: Participants will complete the Generalized Anxiety Disorder 7-item (GAD-7) scale during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks). The survey consisted of 7 questions scored between zero and 21. A score of 5-9 indicates mild severity, 10-14 is moderate, and 15 and greater is considered severe. Data will be presented as the change in anxiety over time compared between groups.
Time Frame: Up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with Generalized Anxiety Disorder 7-item (GAD-7) data available at study time points enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change. Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 26 | 25
score on a scale | 2.0 (5.68) | 1.52 (4.57)

8. Secondary Outcome: Change in Maternal Perceived Stress Over Time
Description: Participants will complete the Perceived Stress Scale 4-item (PSS4) during the second trimester, third trimester, two months postpartum and six months postpartum (up to 50 weeks). The survey consisted of 4 questions scored between zero and 16. Higher scores are correlated with more stress. Data will be presented as the change in stress over time compared between groups.
Time Frame: Up to 50 weeks (enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery))
Population: Overall number of participants analyzed in each Group is based on the number of participants with Perceived Stress Scale 4-item (PSS4) data available at study time points enrollment (up to 31.6 weeks gestation) minus first postpartum visit (2-8.6 weeks after delivery) to determine a change. Disruptions caused by COVID-19 created many challenges in longitudinal data collection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tobacco Intervention | Treatment As Usual
Number analyzed (Participants) | 26 | 24
score on a scale | 0.73 (2.79) | 1.04 (3.17)

ADVERSE EVENTS:
Time Frame: Enrollment (up to 31.6 weeks gestation) through second postpartum visit (20-28.6 weeks after delivery)
Arm/Group | Tobacco Intervention | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 9/38 | 3/38
Other Adverse Events (participants affected / at risk) | 10/38 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobacco Intervention (N=38) | Treatment As Usual (N=38)
Initial or prolonged hospitalization (Pregnancy, puerperium and perinatal conditions) | 5 | 1
Initial or prolonged hospitalization (General disorders) | 4 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobacco Intervention (N=38) | Treatment As Usual (N=38)
Incarceration (Social circumstances) | 4 | 1
Positive response to depression evaluation (General disorders) | 4 | 2
Treatment for dehydration (General disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The B-EPIC study was significantly impacted by the COVID-19 pandemic in terms of recruitment, overall enrollment, and the ability to collect longitudinal data. In spite of the challenges, we were able to enroll 76% of the proposed number of participants in each group. However, power was estimated based on a sample size of 50 per group, and some group comparisons may not have reached significance due to a more limited power given the smaller sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03796208/Prot_SAP_ICF_000.pdf